CLINICAL TRIAL: NCT00614042
Title: A Phase 1/1b Study of TRU-016 in Patients With Previously Treated Chronic Lymphocytic Leukemia or Select Subtypes of Non-Hodgkin's Lymphoma
Brief Title: Phase 1/1b Study of TRU-016 in Patients With Previously Treated CLL or Select Subtypes of Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aptevo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16007
Record Dates: First submitted 2008-01-25; First posted 2008-02-13 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Non-Hodgkin's Lymphoma (NHL)
Keywords: CLL; NHL; TRU-016; chronic lymphocytic leukemia; non-Hodgkin's lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — TRU 016

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Dose escalation and expansion cohorts
  Interventions: Drug: TRU-016 (anti-CD37 protein therapeutic)

INTERVENTIONS:
Drug: TRU-016 (anti-CD37 protein therapeutic) — TRU-016 administered via IV infusion weekly for 8 weeks and then monthly

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of TRU-016 in patients with previously treated chronic lymphocytic leukemia, and to obtain an estimate of clinical activity in patients with CLL and non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
This Phase 1/1b open-label study consists of two parts. The initial portion is a Phase 1 dose-escalation study evaluating the safety and tolerability of TRU-016 administered over a 4-week period to patients with relapsed chronic lymphocytic leukemia (CLL). It will identify the MTD and evaluate the pharmacokinetics and immunogenicity of TRU-016. Upon demonstrating satisfactory safety and tolerability in the Phase 1 portion, a Phase 1b expansion cohort will be enrolled to further characterize the safety of the selected dose from the first stage of the study and safety and to estimate the clinical activity of TRU-016 in patients with treatment-naive CLL, relapsed CLL and non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic lymphocytic lymphoma or small lymphocytic lymphoma (Phase 1) or relapsed/refractory NHL (Phase 1b)
* Previous treatment with at least one fludarabine-containing regimen
* Demonstrate at least one of the following criteria for active disease requiring treatment:

  * a)progressive splenomegaly and/or lymphadenopathy;
  * b)anemia or thrombocytopenia due to bone marrow involvement;
  * c)unintentional weight loss >10% over preceding 6-month period;
  * d) NCI Grade 2 or 3 fatigue;
  * e) fevers >100.5 F or night sweats for > 2 weeks without infection;
  * f) progressive lymphocytosis with increase of >50% over a 2-month period or anticipated doubling time of < 6 months.
* ECOG performance status </= 2
* SGOT, SGPT </= 2.0 x upper limit of normal
* ANC >/= 500/uL
* Platelets >/= 30,000/uL
* Discontinued previous anticancer or investigational therapy for at least 30 days

Exclusion Criteria:

* Treatment with rituximab within 30 days or alemtuzumab(Campath)or radioimmune therapy within 12 weeks
* ANC </= 500/uL
* Platelets </= 30,000/mm3
* Previous or concurrent additional malignancy
* Significant concurrent medical diseases or conditions
* Hepatitis B surface antigen or hepatitis B core antibody positive
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of TRU-016 administered IV in patients with CLL or NHL | 4 weeks after treatment

SECONDARY OUTCOMES:
Preliminary indication of response as defined by NCI 1996 criteria | 3 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Scott Stromatt, MD, Study Director — Aptevo Therapeutics
Locations (7):
- United States (7):
  - For additional information regarding sites for this trial call 919-319-9374, Birmingham, Alabama
  - For additional information regarding sites for this trial call 919-319-9374, Augusta, Georgia
  - For additional information regarding sites for this trial call 919-319-9374, Boston, Massachusetts
  - For additional information regarding sites for this trial call 919-319-9374, Las Vegas, Nevada
  - For additional information regarding sites for this trial call 919-319-9374, Durham, North Carolina
  - For additional information regarding sites for this trial call 919-319-9374, Portland, Oregon
  - For additional information regarding sites for this trial call 919-319-9374, Seattle, Washington

REFERENCES:
- [Result] Pagel JM, Spurgeon SE, Byrd JC, Awan FT, Flinn IW, Lanasa MC, Eisenfeld AJ, Stromatt SC, Gopal AK. Otlertuzumab (TRU-016), an anti-CD37 monospecific ADAPTIR() therapeutic protein, for relapsed or refractory NHL patients. Br J Haematol. 2015 Jan;168(1):38-45. doi: 10.1111/bjh.13099. Epub 2014 Aug 22. PMID 25146490
- [Derived] Byrd JC, Pagel JM, Awan FT, Forero A, Flinn IW, Deauna-Limayo DP, Spurgeon SE, Andritsos LA, Gopal AK, Leonard JP, Eisenfeld AJ, Bannink JE, Stromatt SC, Furman RR. A phase 1 study evaluating the safety and tolerability of otlertuzumab, an anti-CD37 mono-specific ADAPTIR therapeutic protein in chronic lymphocytic leukemia. Blood. 2014 Feb 27;123(9):1302-8. doi: 10.1182/blood-2013-07-512137. Epub 2013 Dec 31. PMID 24381226